CLINICAL TRIAL: NCT01680588
Title: A Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of [18F]NAV4694 PET in the Detection of Beta Amyloid in Subjects With Probable Alzheimer's Disease, Older Healthy Volunteers, and Young Healthy Volunteers
Brief Title: Efficacy and Safety of the PET Imaging Agent [18F]NAV4694 in Subjects With Probable Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV4-01
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]NAV4694 (Experimental): Single intravenous injection of 8.1 millicuries of [18F]NAV4694
  Interventions: Drug: [18F]NAV4694

INTERVENTIONS:
Drug: [18F]NAV4694

SUMMARY:
This is a phase 2, open-label, multiple-center, non-randomized single dose study to assess the safety and efficacy of [18F]NAV4694 PET imaging in detecting beta-amyloid plaque in the brain in subjects with probable AD compared with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* is able to provide informed consent or assent, and exhibits adequate visual, auditory, and communication capabilities to enable compliance with study procedures
* should be able to perform the psychometric testing
* has a modified Hachinski score ((Hachinski, et al., 2012; Rosen, et al., 1980) ≤ 4 at screening
* possesses a general health that permits adequate compliance with all study procedures as ascertained by a detailed review of the medical history, surgical history, laboratory and physical examination findings, which must be performed within 56 days prior to administration of [18F]NAV4694
* informed consent has been signed and dated by the subject and/or the subject's legally authorized representative (LAR; for probable AD subjects)

Healthy Volunteers Only

* is male or female and is between the age of 18 and 40 years (for younger HVs) or 55 to 85 years of age (for older HVs)
* if female does not have childbearing potential: must be confirmed by either: post-menopausal status; or history of surgical sterilization or of hysterectomy
* if female has childbearing potential: must demonstrate a negative serum beta-HCG level at screening and a negative urine pregnancy test on the day of injection (prior to injection) consistent with a non-gravid state and agree to use two acceptable forms of birth control
* has no evidence of cognitive impairment as indicated by a clinical dementia rating (CDR) (Morris, 1993) score of 0 (zero) and a score of ≥ 28 in the Mini-Mental State Examination (MMSE) (Folstein, et al., 1975)
* has MRI brain scan that has been judged as "normal (age-appropriate)" supporting the lack of cerebrovascular disease (e.g., a white matter lesion score of 0, 1, or 2 and a basal ganglia score of 0 to 1 on the ARWMC scale)

Probable Alzheimer's Disease Subjects Only

* is male or female and is ≥ 55 of age, whereby females must be without childbearing potential (confirmed by either:post-menopausal status; or history of surgical sterilization or of hysterectomy)
* presents with positive assessment for dementia of Alzheimer's type in accordance with the DSM-IV-TR and probable AD according to the NINCDS-ADRDA criteria and fulfills none of the exclusion criteria of either
* does not fulfill the International Consensus Criteria (ICC) for probable diffuse Lewy body disease (DLBD), the NINDS-AIREN for probable vascular dementia, or the Neary criteria for frontotemporal dementia (FTD) [Neary et al. 1998]
* has a MMSE score between 16 and 23
* has a CDR (Morris, 1993) score of 1 to 2
* has a Cornell Scale for Depression in Dementia (CSDD; (Alexopoulos, et al., 1988)) score less than or equal to 18 (definite major depression)
* MRI brain scan findings that do not reveal changes indicative of stroke and/or generalized cerebrovascular disease changes (limited to: a white matter lesion score of 0, 1, or 2 and a basal ganglia score of 0 or 1 on the ARWMC scale)
* has a caregiver who is willing and able to attend study visits and perform the psychometric tests requiring the presence of a caregiver

Exclusion Criteria:

* has any contraindication to MRI examination, e.g., metal implants or phobia
* is not able to lie down flat in the MRI and PET scanners
* is scheduled for surgery and/or another invasive procedure within the time period of up to 10 days after [18F]NAV4694 application
* is medically unstable and whose clinical course during the observation period is unpredictable, e.g., subjects within 14 days of myocardial infarction or stroke, unstable subjects with previous surgery (within 7 days), subjects with advanced heart insufficiency (NYHA stage IV), or with acute renal failure
* has a history of exposure to any radiation > 30 mSv in the last year (e.g., occupational, diagnostic imaging, or radiation therapy)
* is receiving drug therapy or other treatment that is known to lead to greatly fluctuating values of the hematological or chemical laboratory parameters or to severe side effects (e.g., chemotherapy)
* has received anti-amyloid immunotherapy
* has been previously enrolled in this study and received [18F]NAV4694 or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening, and/or any radiopharmaceutical within 10 radioactive half-lives prior to [18F]NAV4694 administration
* has a brain tumor or other intracranial lesion, a disturbance of cerebrospinal fluid (CSF) circulation (e.g., normal pressure hydrocephalus) and/or a history of serious head trauma or brain surgery
* has a history, physical, laboratory, or imaging findings indicative of a significant neurological or psychiatric illness (other than AD for the subjects with probable AD)
* has another untreated disease that can cause disturbance of brain function (e.g. vitamin B12 or folic acid deficiency, disturbed thyroid function, anemia)
* has a history of alcohol abuse or drug dependency in the 3 years prior to study entry or is an alcoholic or drug addict as determined by the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
[18F]NAV4694 PET visual assessment by centralized readers | 25 minutes post injection
  To evaluate [18F]NAV4694 PET visual assessment by centralized readers for detection of cerebral beta-amyloid plaque in subjects diagnosed with probable Alzheimer's disease compared with similarly aged and young healthy volunteers.

SECONDARY OUTCOMES:
Assess the incidence of adverse events after a single dose of [18F]NAV4694 | 7 Days
  To assess the incidence of adverse events after a single dose of [18F]NAV4694 PET in individuals diagnosed with probable AD and similarly aged and young healthy volunteers.
Evaluate [18F]NAV4694 PET quantitative assessment | 25 minutes post injection
  To evaluate [18F]NAV4694 PET quantitative assessment, by assessing standard uptake value ratios (SUVR) for detection of cerebral beta-amyloid plaque in subjects diagnosed with probable Alzheimer's disease compared with similarly aged and young healthy volunteers.
Determine correlation of neuro-psychiatric tests with [18F]NAV4694 imaging | 25 minutes post injection
  To determine the correlation of neuro-psychiatric tests with the beta-amyloid plaque burden determined by correlating various baseline neuro-psychiatric test scores with the [18F]NAV4694 PET imaging results in subjects diagnosed with probable AD
Assess changes in laboratory values after a single dose of [18F]NAV4694 | 7 days
  To assess changes in laboratory values after a single dose of [18F]NAV4694 PET in individuals diagnosed with probable AD and similarly aged and young healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Reininger, M.D., PhD, Study Director — Navidea Biopharmaceuticals
Locations (7):
- United States (7):
  - Molecular NeuroImaging, LLC, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Indiana Medical Research, Indianapolis, Indiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Alzheimer's Disease Center, Quincy Medical Center, Quincy, Massachusetts
  - Neurological Associates of Albany, Albany, New York